CLINICAL TRIAL: NCT07287683
Title: Evaluation of Postoperative Pain in Cases Undergoing Cataract Surgery Under Topical Anaesthetic Versus General Anaesthesia
Brief Title: Evaluation of Postoperative Pain in Cases Undergoing Cataract Surgery Under Topical Versus General Anesthesia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, radwa saber, Dr. Radwa Saber, lecturer of Anesthesiology, principal investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0307211
Record Dates: First submitted 2025-09-21; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Topical Anaesthesia; General Anesthetic Drug Adverse Reaction; Cataract
MeSH Terms: conditions — Cataract | interventions — Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group under general anesthesia for cataract surgery (Active Comparator): Patients undergoing cataract surgery will receive general Anaesthesia using intravenous injection and inhalational anaesthetics
  Interventions: Drug: General Anaesthesia group
- Group under topical anaesthesia (Active Comparator): Patients will receive topical anaesthesia for cataract surgery
  Interventions: Drug: Topical Anaesthesia group

INTERVENTIONS:
Drug: Topical Anaesthesia group — This group of patients will only receive topical anaesthesia for Cataract surgery
  Other Names: Topical group
  Arms: Group under topical anaesthesia
Drug: General Anaesthesia group — General Anaesthesia will be given to this group undergoing cataract surgery
  Arms: Group under general anesthesia for cataract surgery

SUMMARY:
Comparison between cataract surgery under local versus general anesthesia regarding postoperative pain, complications and patient satisfaction and need for rescue analgesic intake after surgery The results will be followed up at 24 hrs, 1 week and after one and half month following the surgery.

DETAILED DESCRIPTION:
This prospective randomized controlled study will be carried out on 50 adult patients. Written informed consent will be taken from all prospective cases.

The cases will be selected having (ASA1), (ASA II) or (ASA III) physical status in the age range between 20 and 70 years old with cataract eye disease.

This study will be performed in Alexandria Main University Hospital, Egypt. Patients will be followed up at 24 hours, 1 week, and 6 weeks after surgery.

The following measurements will be recorded

1. Pain will be assessed prior to surgery and after surgery using VAS score at 24 hours, 1 week, and 6 weeks after surgery.
2. Need for analgesic intake after surgery will be assessed for the first 48 hours
3. Complications after surgery as irritation, infection ,and foreign body sensation were assessed
4. Patient satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

- Patients with unilateral cataract planned for surgery under topical or general anesthesia

Exclusion Criteria:

* patients under 20 or over 70 years old Eye infection Patient refusal

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | At 24 hours, one week and 6 weeks following surgery
  Postoperative pain will be assessed using the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
1-complications after surgery 2-Patient satisfaction will be measured using the IOWA Satisfaction with Anaesthesia Scale (ISAS), which ranges from 6 (very satisfied) to 3 or less (dissatisfied). | Up to 6 weeks
  Complications including hypotension, nausea and allergic reaction will be assessed after surgery and 24 hours later. satisfaction assessment will evaluate patient safety, pain control, comfort, nausea, interaction with the surgical team, willingness to repeat the anaesthetic, and relaxation during and after surgery. Patient satisfaction will be recorded at one week and six weeks postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Radwa S Raslan, PHD, Principal Investigator — AMUH
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No